CLINICAL TRIAL: NCT00147498
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Compare 3 Dose Levels Of CP-690,550 Versus Placebo, Administered Orally Twice Daily (BID) For 6 Weeks, In The Treatment Of The Signs And Symptoms Of Subjects With Active Rheumatoid Arthritis
Brief Title: Three Dose Levels of CP-690,550 Monotherapy Versus Placebo, Administered Orally Twice Daily (BID) for 6 Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921019
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis
Keywords: oral JAK inhibitor; clinical trial; joint diseases; anti-Inflammatory agents; rheumatic diseases; DMARD; Antirheumatic Agents; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Joint Diseases; Rheumatic Diseases; Autoimmune Diseases; Immune System Diseases | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 mg BID (Experimental): CP 690,550 5 mg BID
  Interventions: Drug: CP-690,550
- 15 mg BID (Experimental): CP 690,550 15 mg BID
  Interventions: Drug: CP-690,550
- 30 mg BID (Experimental): Oral tablets administered at a dose of 30 mg BID for 6 weeks
  Interventions: Drug: CP-690,550
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CP-690,550 — Oral tablets administered at a dose of 5 mg BID for 6 weeks
  Arms: 5 mg BID
Drug: CP-690,550 — Oral tablets administered at a dose of 15 mg BID for 6 weeks
  Arms: 15 mg BID
Drug: CP-690,550 — 30 mg BID for 6 weeks
  Arms: 30 mg BID
Other: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
The study's objective is to compare the efficacy of 3 dose levels of oral CP-690,550 monotherapy (5 mg, 15 mg, and 30 mg twice daily [BID]) versus placebo administered over 6 weeks for the treatment of the signs and symptoms of subjects with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* The subject has a history of inadequate response to at least 1, but no more than 4, of the following DMARDs: sulfasalazine, injectable gold, methotrexate, leflunomide, cyclosporine, or a thiopurine derivative (azathioprine or 6-mercaptopurine)

Exclusion Criteria:

* Current Therapy With Any DMARD Or Biologic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- United States (22):
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Concord, New Hampshire
  - Pfizer Investigational Site, Plainview, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Ducansville, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Pfizer Investigational Site, Ghent, Belgium
- Brazil (3):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (5):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hildesheim
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Neubrandenburg
  - Pfizer Investigational Site, Wiesbaden
- Italy (3):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Pavia
- Mexico (5):
  - Pfizer Investigational Site, Aguascalientes, Aguascalientes
  - Pfizer Investigational Site, México, D.f.
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Tlalpan Seccion 16, Mexico City
  - Pfizer Investigational Site, San Luis Potosí City, San Luis Potosí
- Slovakia (3):
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Žilina
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Guadalajara, Guadalajara
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Mariette X, Chen C, Biswas P, Kwok K, Boy MG. Lymphoma in the Tofacitinib Rheumatoid Arthritis Clinical Development Program. Arthritis Care Res (Hoboken). 2018 May;70(5):685-694. doi: 10.1002/acr.23421. Epub 2018 Apr 2. PMID 28941219
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Kremer JM, Bloom BJ, Breedveld FC, Coombs JH, Fletcher MP, Gruben D, Krishnaswami S, Burgos-Vargas R, Wilkinson B, Zerbini CA, Zwillich SH. The safety and efficacy of a JAK inhibitor in patients with active rheumatoid arthritis: Results of a double-blind, placebo-controlled phase IIa trial of three dosage levels of CP-690,550 versus placebo. Arthritis Rheum. 2009 Jul;60(7):1895-905. doi: 10.1002/art.24567. PMID 19565475
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921019&StudyName=Three%20Dose%20Levels%20of%20CP-690%2C550%20Monotherapy%20Versus%20Placebo%2C%20Administered%20Orally%20Twice%20Daily%20%28BID%29%20for%206%20Weeks

RESULTS

PARTICIPANT FLOW:
Groups:
- CP 690,550 5 mg: CP-690,550 tablets equivalent to CP-690,550 5 milligram (mg) orally twice daily for 6 weeks.
- CP-690,550 15 mg: CP-690,550 tablets equivalent to CP-690,550 15 mg orally twice daily for 6 weeks.
- CP-690,550 30 mg: CP-690,550 tablets equivalent to CP-690,550 30 mg orally twice daily for 6 weeks.
- Placebo: Placebo matched to CP-690,550 tablets orally twice daily for 6 weeks.
Period: Overall Study
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Started | 61 | 69 | 69 | 65
Completed | 58 | 60 | 52 | 48
Not Completed | 3 | 9 | 17 | 17
Not completed — Adverse Event | 1 | 6 | 7 | 3
Not completed — Lack of Efficacy | 1 | 1 | 1 | 8
Not completed — Laboratory abnormality | 0 | 0 | 2 | 0
Not completed — Participant defaulted | 0 | 1 | 4 | 3
Not completed — Other | 1 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo | Total
Number analyzed (Participants) | 61 | 69 | 69 | 65 | 264
Age Continuous [Mean (Standard Deviation); unit: years] | 47.9 (10.8) | 51.8 (13.0) | 51.1 (10.6) | 51.3 (12.1) | 50.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 58 | 60 | 55 | 226
  Male | 8 | 11 | 9 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 6
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joints count (TJC); >= 20% improvement in swollen joints count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 6
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 69 | 65
percentage of participants | 70.49 | 81.16 | 76.81 | 29.23

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: >=20% improvement in TJC; >= 20% improvement in SJC; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, and 8
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Missing data were imputed using Last Observation Carried Forward (LOCF) at Week 1, 2, and 4. Here 'n' is number of participants evaluable at specific time points for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 69 | 65
percentage of participants
  Week 1 (n=61,69,69,65) | 27.87 | 43.48 | 56.52 | 12.31
  Week 2 (n=61,69,69,65) | 50.82 | 71.01 | 68.12 | 20.00
  Week 4 (n=61,69,69,65) | 63.93 | 75.36 | 75.36 | 30.77
  Week 8 (n=56,56,51,45) | 50.00 | 66.07 | 70.59 | 28.89

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >= 50% improvement in TJC or SJC and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, 6, and 8
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Missing data were imputed using Last Observation Carried Forward (LOCF) at Week 1, 2, 4, and 6. Here 'n' is number of participants evaluable at specific time points for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 69 | 65
percentage of participants
  Week 1 (n= 61,69,69,65) | 6.56 | 8.70 | 18.84 | 3.08
  Week 2 (n= 61,69,69,65) | 9.84 | 23.19 | 28.99 | 3.08
  Week 4 (n= 61,69,69,65) | 32.79 | 42.03 | 42.03 | 6.15
  Week 6 (n= 61,69,69,65) | 32.79 | 53.62 | 50.72 | 6.15
  Week 8 (n=56,56,51,45) | 17.86 | 30.36 | 45.10 | 13.33

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >= 70% improvement in TJC or SJC and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, 6, and 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 69 | 65
percentage of participants
  Week 1 (n= 61,69,69,65) | 1.64 | 4.35 | 4.35 | 0.00
  Week 2 (n= 61,69,69,65) | 4.92 | 4.35 | 10.14 | 1.54
  Week 4 (n= 61,69,69,65) | 9.84 | 17.39 | 21.74 | 1.54
  Week 6 (n= 61,69,69,65) | 13.11 | 21.74 | 27.54 | 3.08
  Week 8 (n=56,56,51,45) | 8.93 | 14.29 | 27.45 | 8.89

5. Secondary Outcome: Area Under the Numeric Index of American College of Rheumatology Response (ACR-n) Curve
Description: ACR-n: calculated by taking the lowest percentage improvement in (1) SJC or (2) TJC or (3) the median of the remaining 5 components of the ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening. The area under the curve (AUC) for ACR-n is the measure of the AUC of the mean change from baseline in ACR-n. The trapezoidal rule was used to compute the AUC.
Time Frame: Baseline up to Week 6
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale*weeks
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 59 | 69 | 66 | 62
units on a scale*weeks | 857.50 (1151.36) | 1086.90 (1664.77) | 1211.93 (2107.65) | -546.41 (1721.78)

6. Secondary Outcome: Tender Joints Count (TJC)
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure and 'n' is number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 68 | 65
tender joints
  Baseline (n=61,69,68,65) | 32.37 (1.588) | 26.98 (1.485) | 29.52 (1.499) | 30.61 (1.529)
  Week 1 (n=60,68,66,59) | 23.49 (1.597) | 16.62 (1.492) | 15.75 (1.511) | 27.39 (1.576)
  Week 2 (n=57,66,65,60) | 18.90 (1.622) | 12.72 (1.505) | 13.51 (1.519) | 24.71 (1.572)
  Week 4 (n=56,58,59,49) | 15.33 (1.628) | 9.97 (1.562) | 10.17 (1.562) | 19.78 (1.670)
  Week 6 (n=56,59,53,50) | 12.21 (1.630) | 8.58 (1.556) | 7.41 (1.612) | 19.81 (1.661)
  Week 8 (n=57,56,52,45) | 16.32 (1.62) | 11.50 (1.58) | 11.21 (1.62) | 20.37 (1.71)

7. Secondary Outcome: Change From Baseline in Tender Joints Count (TJC) at Week 1, 2, 4, 6 and 8
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from baseline indicated an improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 60 | 68 | 65 | 59
tender joints
  Change at Week 1 (n=60,68,65,59) | -7.06 (1.435) | -11.70 (1.338) | -14.14 (1.362) | -2.74 (1.417)
  Change at Week 2 (n=57,66,65,60) | -11.68 (1.459) | -15.66 (1.350) | -15.78 (1.365) | -5.13 (1.416)
  Change at Week 4 (n=56,58,58,49) | -15.23 (1.465) | -18.33 (1.403) | -18.66 (1.413) | -10.09 (1.508)
  Change at Week 6 (n=56,59,52,50) | -18.35 (1.466) | -19.81 (1.398) | -21.37 (1.461) | -9.69 (1.500)
  Change at Week 8 (n=57,56,52,45) | -14.26 (1.46) | -16.89 (1.42) | -17.78 (1.46) | -9.34 (1.55)

8. Secondary Outcome: Swollen Joints Count (SJC)
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 68 | 65
swollen joints
  Baseline (n=61,69,68,65) | 21.33 (1.052) | 16.42 (0.984) | 19.53 (0.993) | 19.97 (1.013)
  Week 1 (n=60,68,66,59) | 14.77 (1.058) | 9.90 (0.989) | 10.18 (1.001) | 16.46 (1.044)
  Week 2 (n=57,66,65,60) | 12.04 (1.074) | 6.84 (0.997) | 7.99 (1.006) | 14.30 (1.041)
  Week 4 (n=56,58,59,49) | 8.83 (1.079) | 5.95 (1.035) | 6.42 (1.035) | 11.78 (1.107)
  Week 6 (n=56,59,53,50) | 7.74 (1.080) | 4.93 (1.031) | 4.95 (1.069) | 11.15 (1.101)
  Week 8 (n=57,56,52,45) | 10.31 (1.07) | 6.02 (1.05) | 6.77 (1.08) | 12.36 (1.14)

9. Secondary Outcome: Change From Baseline in Swollen Joints Count (SJC) at Week 1, 2, 4, 6 and 8
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 60 | 68 | 65 | 60
swollen joints
  Change at Week 1 (n=60,68,65,59) | -5.02 (0.913) | -8.20 (0.855) | -9.00 (0.866) | -3.19 (0.900)
  Change at Week 2 (n=57,66,65,60) | -7.83 (0.927) | -11.33 (0.863) | -11.11 (0.868) | -5.23 (0.900)
  Change at Week 4 (n=56,58,58,49) | -11.03 (0.930) | -12.10 (0.894) | -12.58 (0.897) | -7.73 (0.954)
  Change at Week 6 (n=56,59,52,50) | -12.10 (0.931) | -13.13 (0.891) | -13.91 (0.925) | -8.06 (0.950)
  Change at Week 8 (n=57,56,52,45) | -9.54 (0.93) | -12.02 (0.90) | -12.14 (0.93) | -7.00 (0.98)

10. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 millimeter (mm) Visual Analog Scale (VAS) where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 58 | 67 | 65 | 63
mm
  Baseline (n=57,67,65,63) | 71.03 (3.126) | 69.37 (2.887) | 63.99 (2.941) | 65.73 (2.985)
  Week 1 (n=58,67,64,58) | 49.89 (3.111) | 45.36 (2.889) | 39.79 (2.958) | 61.48 (3.076)
  Week 2 (n=55,65,62,60) | 46.18 (3.171) | 41.09 (2.917) | 32.09 (2.992) | 58.02 (3.046)
  Week 4 (n=56,58,58,48) | 38.67 (3.146) | 29.53 (3.033) | 26.16 (3.062) | 52.55 (3.294)
  Week 6 (n=55,59,52,49) | 37.11 (3.165) | 28.82 (3.018) | 24.52 (3.180) | 50.04 (3.273)
  Week 8 (n=57,57,50,45) | 40.29 (3.13) | 37.56 (3.05) | 30.63 (3.23) | 50.76 (3.37)

11. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) of Arthritis at Week 1, 2, 4, 6 and 8
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 56 | 66 | 62 | 59
mm
  Change at Week 1 (n=56,66,62,57) | -17.98 (3.121) | -21.56 (2.859) | -26.16 (2.948) | -5.18 (3.022)
  Change at Week 2 (n=53,63,60,59) | -22.06 (3.184) | -25.71 (2.900) | -33.33 (2.984) | -8.14 (2.998)
  Change at Week 4 (n=53,57,55,47) | -30.23 (3.176) | -37.35 (3.001) | -38.71 (3.072) | -13.17 (3.238)
  Change at Week 6 (n=52,57,49,48) | -31.64 (3.203) | -37.78 (3.005) | -40.50 (3.191) | -15.06 (3.219)
  Change at Week 8 (n=53,55,48,45) | -27.83 (3.18) | -28.79 (3.04) | -34.30 (3.21) | -14.96 (3.28)

12. Secondary Outcome: Physician Global Assessment of Arthritis
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 60 | 69 | 66 | 64
mm
  Baseline (n=60,69,66,64) | 69.39 (2.566) | 64.11 (2.388) | 66.65 (2.436) | 67.75 (2.471)
  Week 1 (n=60,67,64,58) | 49.85 (2.568) | 37.80 (2.417) | 36.30 (2.464) | 55.54 (2.575)
  Week 2 (n=57,66,65,60) | 41.65 (2.618) | 29.54 (2.430) | 32.24 (2.453) | 52.76 (2.546)
  Week 4 (n=56,58,59,49) | 34.18 (2.631) | 27.45 (2.547) | 23.91 (2.540) | 46.01 (2.746)
  Week 6 (n=55,58,53,50) | 31.42 (2.651) | 22.22 (2.549) | 19.26 (2.643) | 46.52 (2.727)
  Week 8 (n=57,57,52,45) | 39.10 (2.62) | 30.78 (2.57) | 26.24 (2.66) | 42.04 (2.84)

13. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis at Week 1, 2, 4, 6 and 8
Description: as for outcome 12
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 59 | 67 | 63 | 59
mm
  Change at Week 1 (n=59,67,62,57) | -17.13 (2.626) | -28.25 (2.445) | -30.89 (2.534) | -12.25 (2.636)
  Change at Week 2 (n=56,66,63,59) | -25.43 (2.675) | -36.60 (2.456) | -34.56 (2.525) | -14.29 (2.611)
  Change at Week 4 (n=55,58,56,48) | -33.29 (2.686) | -38.44 (2.563) | -42.65 (2.627) | -20.91 (2.803)
  Change at Week 6 (n=55,58,50,49) | -35.97 (2.690) | -43.69 (2.566) | -46.70 (2.730) | -19.87 (2.786)
  Change at Week 8 (n=56,57,50,45) | -29.19 (2.67) | -35.11 (2.58) | -39.81 (2.73) | -24.78 (2.87)

14. Secondary Outcome: Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 59 | 68 | 66 | 64
mm
  Baseline (n=59,68,66,64) | 69.46 (3.112) | 67.47 (2.894) | 68.13 (2.936) | 64.17 (2.980)
  Week 1 (n=59,68,65,59) | 51.76 (3.114) | 46.11 (2.897) | 37.71 (2.953) | 62.51 (3.072)
  Week 2 (n=57,65,65,60) | 45.59 (3.154) | 40.14 (2.940) | 30.83 (2.956) | 60.65 (3.062)
  Week 4 (n=57,58,59,49) | 37.77 (3.150) | 30.42 (3.057) | 26.76 (3.053) | 56.96 (3.287)
  Week 6 (n=55,59,53,50) | 35.57 (3.191) | 28.35 (3.043) | 23.39 (3.169) | 52.75 (3.266)
  Week 8 (n=57,57,52,45) | 42.44 (3.15) | 37.62 (3.08) | 31.12 (3.19) | 49.06 (3.39)

15. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritis Pain at Week 1, 2, 4, 6 and 8
Description: as for outcome 14
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 57 | 67 | 63 | 59
mm
  Change at Week 1 (n=57,67,63,58) | -15.01 (3.102) | -19.74 (2.843) | -29.66 (2.932) | -3.30 (3.027)
  Change at Week 2 (n=55,65,63,59) | -21.44 (3.142) | -26.10 (2.870) | -35.85 (2.936) | -4.79 (3.027)
  Change at Week 4 (n=55,57,56,48) | -29.27 (3.137) | -35.47 (2.996) | -40.10 (3.050) | -8.40 (3.242)
  Change at Week 6 (n=54,58,51,49) | -31.42 (3.159) | -37.67 (2.983) | -42.89 (3.144) | -12.26 (3.223)
  Change at Week 8 (n=55,56,51,45) | -24.90 (3.14) | -28.70 (3.02) | -35.35 (3.15) | -16.28 (3.31)

16. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 60 | 69 | 67 | 62
units on a scale
  Baseline (n=60,69,67,62) | 1.75 (0.086) | 1.66 (0.080) | 1.61 (0.081) | 1.71 (0.083)
  Week 1 (n=60,68,65,58) | 1.46 (0.086) | 1.37 (0.080) | 1.19 (0.082) | 1.63 (0.084)
  Week 2 (n=57,66,64,60) | 1.32 (0.087) | 1.17 (0.081) | 1.06 (0.082) | 1.53 (0.084)
  Week 4 (n=57,57,59,47) | 1.17 (0.087) | 1.07 (0.083) | 0.92 (0.083) | 1.54 (0.088)
  Week 6 (n=54,59,53,50) | 1.12 (0.088) | 0.95 (0.082) | 0.86 (0.084) | 1.47 (0.087)
  Week 8 (n=57,56,52,45) | 1.30 (0.09) | 1.06 (0.08) | 0.92 (0.08) | 1.52 (0.09)

17. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 1, 2, 4, 6 and 8
Description: as for outcome 16
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 59 | 68 | 64 | 57
units on a scale
  Change at Week 1 (n=59,68,64,55) | -0.25 (0.066) | -0.30 (0.061) | -0.44 (0.063) | -0.05 (0.067)
  Change at Week 2 (n=56,66,63,57) | -0.39 (0.067) | -0.50 (0.062) | -0.56 (0.063) | -0.15 (0.067)
  Change at Week 4 (n=56,57,57,44) | -0.55 (0.067) | -0.60 (0.064) | -0.69 (0.065) | -0.13 (0.071)
  Change at Week 6 (n=55,59,51,47) | -0.60 (0.068) | -0.72 (0.063) | -0.74 (0.067) | -0.20 (0.070)
  Change at Week 8 (n=56,56,51,43) | -0.43 (0.07) | -0.60 (0.06) | -0.70 (0.07) | -0.17 (0.07)

18. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is 0 milligram per liter (mg/L) to 100 mg/L. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 50 | 57 | 58 | 53
mg/L
  Baseline (n=50,57,58,53) | 31.25 (35.00) | 25.47 (31.06) | 28.10 (28.43) | 22.28 (18.52)
  Week 1 (n=50,55,55,49) | 15.98 (16.72) | 7.57 (9.79) | 7.57 (11.32) | 25.40 (30.04)
  Week 2 (n=46,53,53,48) | 13.18 (12.97) | 7.25 (11.83) | 6.50 (14.81) | 24.41 (21.38)
  Week 4 (n=46,49,47,39) | 11.83 (11.10) | 5.17 (6.72) | 5.88 (10.98) | 22.26 (21.07)
  Week 6 (n=45,49,41,41) | 12.57 (21.01) | 6.59 (16.37) | 6.08 (11.80) | 22.94 (20.79)
  Week 8 (n=45,45,41,37) | 23.37 (22.72) | 12.06 (12.20) | 13.95 (14.68) | 23.64 (29.47)

19. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 1, 2, 4, 6 and 8
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is 0 mg/L to 100 mg/L. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 50 | 54 | 55 | 48
mg/L
  Change at Week 1 (n=50,54,55,48) | -15.28 (26.65) | -18.29 (28.98) | -21.38 (25.56) | -0.24 (15.40)
  Change at Week 2 (n=46,52,53,48) | -16.74 (32.94) | -18.89 (31.87) | -23.06 (31.49) | 1.79 (15.56)
  Change at Week 4 (n=46,49,47,39) | -17.76 (33.31) | -22.02 (31.29) | -20.70 (25.69) | -0.67 (19.17)
  Change at Week 6 (n=45,49,41,41) | -17.83 (35.92) | -18.08 (25.99) | -17.58 (24.76) | 0.67 (16.81)
  Change at Week 8 (n=45,45,41,37) | -7.06 (35.75) | -13.24 (27.69) | -11.81 (29.46) | 1.32 (27.26)

20. Secondary Outcome: Disease Activity Score Using 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score ranging 0 to 9.4; higher scores indicated greater affectation due to disease activity. DAS 28-3 (CRP) less than or equal to (<=) 3.2 implied low disease activity and greater than (>) 3.2 to 5.1 implied moderate to high disease activity, and less than (<) 2.6 = remission.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 50 | 57 | 56 | 51
units on a scale
  Baseline (n=50,57,56,51) | 6.17 (0.89) | 5.69 (0.92) | 5.91 (0.91) | 6.00 (0.90)
  Week 1 (n=49,54,54,47) | 5.29 (1.08) | 4.42 (1.12) | 4.28 (1.21) | 5.66 (1.10)
  Week 2 (n=46,53,51,48) | 4.93 (1.08) | 3.80 (1.17) | 3.90 (1.17) | 5.37 (1.15)
  Week 4 (n=46,49,47,39) | 4.44 (1.20) | 3.56 (1.12) | 3.46 (1.33) | 4.91 (1.22)
  Week 6 (n=45,49,40,41) | 4.18 (1.29) | 3.42 (1.16) | 3.10 (1.17) | 4.78 (1.05)
  Week 8 (n=45,44,41,36) | 4.75 (1.37) | 4.08 (1.32) | 3.93 (1.38) | 5.02 (1.10)

21. Secondary Outcome: Change From Baseline in Disease Activity Score Using 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Week 1, 2, 4, 6, and 8
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score ranging 0 to 9.4; higher scores indicated greater affectation due to disease activity. DAS 28-3 (CRP) <=3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and <2.6 = remission.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: FAS included all participants who were randomized to study treatment. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants who were evaluable for a particular time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 49 | 53 | 52 | 46
units on a scale
  Change at Week 1 (n=49,53,52,45) | -0.84 (0.74) | -1.28 (0.99) | -1.65 (0.99) | -0.39 (0.86)
  Change at Week 2 (n=46,52,50,46) | -1.19 (0.89) | -1.91 (1.23) | -2.05 (1.25) | -0.59 (0.98)
  Change at Week 4 (n=46,49,46,37) | -1.64 (1.16) | -2.18 (1.25) | -2.47 (1.39) | -1.04 (1.04)
  Change at Week 6 (n=45,49,39,39) | -1.99 (1.28) | -2.28 (1.33) | -2.73 (1.32) | -1.20 (1.17)
  Change at Week 8 (n=45,44,41,35) | -1.36 (1.32) | -1.60 (1.32) | -1.99 (1.38) | -0.89 (1.07)

22. Secondary Outcome: Number of Participants With Categorization of Disease Improvement Based on DAS28-3 (CRP)
Description: Disease improvement was classified as good, moderate, and no change based on improvement in DAS 28-3 (CRP) from baseline and present DAS 28-3 (CRP) score. Good: an improvement from baseline of >1.2 and a present score of <=3.2; none: an improvement of <=0.6 or >0.6 to <=1.2 with a present score of >5.1; remaining participants were classified as having moderate improvement. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Baseline, Week 1, 2, 4, 6, and 8
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Number analyzed (Participants) | 49 | 53 | 52 | 46
participants
  Week 1, No Change (n=49,53,52,45) | 31 | 25 | 17 | 35
  Week 1, Good (n=49,53,52,45) | 0 | 0 | 0 | 0
  Week 1, Moderate (n=49,53,52,45) | 18 | 28 | 35 | 10
  Week 2, No Change (n=46,52,50,46) | 20 | 13 | 12 | 33
  Week 2, Good (n=46,52,50,46) | 0 | 0 | 0 | 0
  Week 2, Moderate (n=46,52,50,46) | 26 | 39 | 38 | 13
  Week 4, No Change (n=46,49,46,37) | 14 | 7 | 8 | 22
  Week 4, Good (n=46,49,46,37) | 0 | 0 | 0 | 0
  Week 4, Moderate (n=46,49,46,37) | 32 | 42 | 38 | 15
  Week 6, No Change (n=45,49,39,39) | 11 | 8 | 3 | 20
  Week 6, Good (n=45,49,39,39) | 0 | 0 | 0 | 0
  Week 6, Moderate (n=45,49,39,39) | 34 | 41 | 36 | 19
  Week 8, No Change (n=45,44,41,35) | 21 | 16 | 11 | 24
  Week 8, Good (n=45,44,41,35) | 0 | 0 | 0 | 0
  Week 8, Moderate (n=45,44,41,35) | 24 | 28 | 30 | 11

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP 690,550 5 mg | CP-690,550 15 mg | CP-690,550 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/61 | 5/69 | 3/69 | 1/65
Other Adverse Events (participants affected / at risk) | 34/61 | 38/69 | 46/69 | 37/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP 690,550 5 mg (N=61) | CP-690,550 15 mg (N=69) | CP-690,550 30 mg (N=69) | Placebo (N=65)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Whipple's disease (Infections and infestations) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP 690,550 5 mg (N=61) | CP-690,550 15 mg (N=69) | CP-690,550 30 mg (N=69) | Placebo (N=65)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 7 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 6 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 2
Fatigue (General disorders) | 1 | 2 | 1 | 0
Malaise (General disorders) | 0 | 1 | 3 | 0
Oedema peripheral (General disorders) | 3 | 1 | 3 | 2
Gastroenteritis (Infections and infestations) | 2 | 2 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 2 | 2 | 0
Influenza (Infections and infestations) | 3 | 2 | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3
Tinea pedis (Infections and infestations) | 0 | 3 | 1 | 0
Tinea versicolour (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 5 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 3 | 1
Headache (Nervous system disorders) | 10 | 8 | 17 | 6
Somnolence (Nervous system disorders) | 0 | 2 | 2 | 1
Leukocyturia (Renal and urinary disorders) | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 1
Hypertension (Vascular disorders) | 1 | 2 | 3 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.